CLINICAL TRIAL: NCT03868982
Title: Lung Protection in Acute Respiratory Distress Syndrome Using Neurally Adjusted Ventilatory Assist
Brief Title: Lung Protection in ARDS Using Neurally Adjusted Ventilatory Assist
Acronym: NAVA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fu Jen Catholic University (Other)
Responsible Party: Principal Investigator, Ke-Yun, Chao, Group leader of Respiratory Therapists, Fu Jen Catholic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PL-201808006-V
Record Dates: First submitted 2019-03-04; First posted 2019-03-11 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-02

CONDITIONS: ARDS, Human; Mechanical Ventilation Pressure High
Keywords: acute respiratory distress syndrome; neurally adjusted ventilatory assist; lung protective strategy
MeSH Terms: conditions — Respiratory Distress Syndrome | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Intervention Model Description: Fifty participant with ARDS according to the Berlin Definition will enroll to this study. Participants studied twice daily with collection of data and blood tests.
Who Masked: Participant
Masking Description: Participants will be randomized into study group or control group, and which is single blind processes to participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAVA group (Experimental): Participent in this group will received NAVA for two days
  Interventions: Device: Neurally adjusted ventilatory assist
- Control group (No Intervention): Participent in this group will received standard care

INTERVENTIONS:
Device: Neurally adjusted ventilatory assist — NAVA uses the diaphragm activity to deliver mechanical ventilation
  Arms: NAVA group

SUMMARY:
The aim of this study is to investigate the use neurally adjusted ventilatory assist (NAVA) as lung protective strategy in patients with acute respiratory distress syndrome (ARDS).

DETAILED DESCRIPTION:
Background： Acute respiratory distress syndrome (ARDS) should ventilated with a tidal volume of 4-6 ml/kg according to the ARDSnet recommendations. Due to the lack of clinical evidence of the potential role of neurally adjusted ventilatory assist (NAVA) in ARDS, investigators would like to conduct a study comparing the two modes from a lung protective point of view. Investigators believe it may have a great value in defining guidelines for improved lung protection.

Study Design： This is a prospective, pilot-randomized controlled trial n a single intensive care unit from one hospital. The study is expected to close the case a year (2018.08.01-2019.07.31).

Methods： Fifty patients with ARDS according to the Berlin Definition will enroll to this study. Patients are randomized after fulfilling inclusion and none of the exclusion criteria (25 participants will divide into study group and the other 25 participants will be control group). Patients are studied twice daily with collection of data and blood tests. All data are collected and analysis.

Effect： Tidal volumes in ARDS patients ventilated with NAVA will show tidal volumes clearly within the safe range. ARDS patients on NAVA mode will show improvements in oxygenation, gas distribution and inflammatory markers while requiring less sedatives and hemodynamic support.

Key words： Acute respiratory distress syndrome; neurally adjusted ventilatory assist; lung protective strategy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ARDS by Berlin definition
* P/F ratio between 100-300
* Completed the case enrollement within 48 hours

Exclusion Criteria:

* Less than 18 years old
* Pregnancy
* Participants with tracheostomy
* Unable to insert the NG-tube

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-18 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
PaO2/FiO2 ratio | 2 days
  PaO2 is a data from ABG; FiO2 is the data of ventilator deliver oxygen

SECONDARY OUTCOMES:
PaCO2 | 2 days
  PaCO2 is a data from ABG, represent in mmHg
Tidal volume | 2 days
  Tidal volume is represent in ml
Mechanical ventilation days | 3 months
  MV days
Length of hospital stay | 3 months
  hospital days
Length of intensive care unit stay | 3 months
  ICU days

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Lun Liu, MD, Principal Investigator — Department of Emergency and Critical Care Medicine, Fu Jen Catholic University Hospital, Fu Jen Catholic University
Locations (1):
- Fu Jen Catholic University Hospital, Fu Jen Catholic University, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Navalesi P, Colombo D, Della Corte F. NAVA ventilation. Minerva Anestesiol. 2010 May;76(5):346-52. PMID 20395897
- [Background] Bourenne J, Guervilly C, Mechati M, Hraiech S, Fraisse M, Bisbal M, Roch A, Forel JM, Papazian L, Gainnier M. Variability of reverse triggering in deeply sedated ARDS patients. Intensive Care Med. 2019 May;45(5):725-726. doi: 10.1007/s00134-018-5500-6. Epub 2019 Feb 28. No abstract available. PMID 30820583
- [Background] Assy J, Mauriat P, Tafer N, Soulier S, El Rassi I. Neurally adjusted ventilatory assist for children on veno-venous ECMO. J Artif Organs. 2019 Jun;22(2):118-125. doi: 10.1007/s10047-018-01087-y. Epub 2019 Jan 4. PMID 30610519